CLINICAL TRIAL: NCT06861712
Title: Neoadjuvant Chemoimmunotherapy With or Without SBRT Followed by Surgery for Locoregionally Advanced Squamous Cell Carcinoma of the Oral Cavity and Oropharynx: A Phase II Randomized Trial
Brief Title: Chemoimmunotherapy With or Without SBRT Before Surgery for Locally Advanced Oral and Oropharyngeal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Hospital of Stomatology, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Fang-Yun Xie, Principal Investigator, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2024-858-01
Record Dates: First submitted 2025-02-24; First posted 2025-03-06 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Oral Squamous Cell Carcinoma (OSCC); Oropharyngeal Squamous Cell Carcinoma (SCC); Stereotactic Body Radiation Therapy (SBRT)
Keywords: Oral Squamous Cell Carcinoma (OSCC); Oropharyngeal Squamous Cell Carcinoma (SCC); Stereotactic Body Radiation Therapy (SBRT); Toripalimab; Phase II Clinical Trial
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Docetaxel; Cisplatin; toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): The experimental group will first receive SBRT (Stereotactic Body Radiotherapy) for the primary tumor and positive lymph nodes (prescribed dose: 6 Gy × 3 fractions, once every other day). One to two weeks after SBRT, they will receive 240 mg of Toripalimab (provided) + 75 mg/m² of Docetaxel + 75 mg/m² of Cisplatin, administered every 3 weeks for 3 cycles.
  Interventions: Radiation: SBRT; Drug: Docetaxel, Cisplatin, Toripalimab; Procedure: Radical resection surgery; Radiation: IMRT ± chemotherapy/toripalimab
- Control Group (Active Comparator): The control group will directly receive 240 mg of Toripalimab + 75 mg/m² of Docetaxel + 75 mg/m² of Cisplatin, administered every 3 weeks for 3 cycles.
  Interventions: Drug: Docetaxel, Cisplatin, Toripalimab; Procedure: Radical resection surgery; Radiation: IMRT ± chemotherapy/toripalimab

INTERVENTIONS:
Radiation: SBRT — The experimental group will first receive SBRT (Stereotactic Body Radiotherapy) for the primary tumor and positive lymph nodes (prescribed dose: 6 Gy × 3 fractions, once every other day).
  Arms: Experimental Group
Drug: Docetaxel, Cisplatin, Toripalimab — Toripalimab 240mg (free medicine) + Docetaxel 75mg/m2 + Cisplatin 75mg/m2, q3w for 3 courses
  Other Names: Neoadjuvant Chemoimmunotherapy
Procedure: Radical resection surgery — Radical resection surgery
Radiation: IMRT ± chemotherapy/toripalimab — According to the preoperative staging and postoperative pathological characteristics, all patients will receive postoperative radiotherapy with or without cisplatin-based chemotherapy. Additionally, patients can choose whether to continue maintenance therapy with toripalimab after surgery.

SUMMARY:
In this study, participants will be randomly assigned to either the experimental group or the control group. The experimental group will first receive SBRT (6Gy*3 fractions) to treat the primary tumor and metastatic lymph nodes. This will be followed by a combination of Toripalimab, Docetaxel, and Cisplatin for three cycles, every three weeks. The control group will receive the same combination of Toripalimab, Docetaxel, and Cisplatin for three cycles, every three weeks, but without SBRT. After the final round of chemotherapy, all participants will have imaging scans and, three weeks later, undergo surgery. After surgery, they may also receive additional radiotherapy with or without chemotherapy. Patients can also choose whether to continue treatment with Toripalimab after surgery.

DETAILED DESCRIPTION:
Participants will be randomly assigned to the experimental group and the control group. The experimental group will first receive SBRT (Stereotactic Body Radiotherapy) for the primary tumor and positive lymph nodes (prescribed dose: 6 Gy × 3 fractions, once every other day). One to two weeks after SBRT, they will receive 240 mg of Toripalimab + 75 mg/m² of Docetaxel + 75 mg/m² of Cisplatin, administered every 3 weeks for 3 cycles. The control group will receive 240 mg of Toripalimab + 75 mg/m² of Docetaxel + 75 mg/m² of Cisplatin, administered every 3 weeks for 3 cycles. Both groups will undergo imaging assessment 2 weeks after the final chemotherapy cycle. Three weeks after the last chemotherapy cycle, participants will receive curative surgery. Postoperative adjuvant radiotherapy ± chemotherapy will be administered according to preoperative staging and postoperative pathological characteristics. Patients may also choose to continue maintenance treatment with Toripalimab after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Oral/oropharyngeal squamous cell carcinoma confirmed by histology and/or cytology.
2. Clinical stage: resectable oral/oropharyngeal squamous cell carcinoma stage III-IVa (AJCC 8th edition)
3. Age: 18-65 years old.
4. According to the Eastern Cooperative Oncology Group (ECOG) criteria (performance status score of 0 or 1).
5. Good organ function:

   A. Hematology: WBC ≥ 4000/μL, neutrophil ≥ 2.000/μL, hemoglobin ≥ 9g/dL, platelet ≥ 100000/μL; B. Liver function: bilirubin ≤ 1.5 times the upper limit of normal (ULN) (patients with known Gilbert's disease and serum bilirubin level ≤ 3 times ULN can be included), AST and ALT ≤ 3 times, and alkaline phosphatase ≤ 3 times ULN; albumin ≥ 3g/dL; C. International normalized ratio (INR) or prothrombin time (PT) or activated partial thromboplastin time (aPTT) ≤ 1.5 times; D. Renal function: serum creatinine ≤ 1.5 times ULN or creatinine clearance ≥ 60mL/min according to the Cockcroft-Gault formula.
6. Expected survival ≥ 3 months.
7. The patient has signed an informed consent form and is willing and able to comply with the study visits, treatment plans, laboratory tests and other study procedures.
8. Women of childbearing potential must have a negative urine or serum pregnancy test within 7 days before enrollment and must agree to take effective contraceptive measures during the study and for at least 60 days after the last dose (including chemotherapy drugs and Teplizumab).
9. If the female partner of the male subject is still of childbearing potential, the male subject must agree to take effective contraceptive measures during the study and for at least 60 days after the last dose.

Exclusion Criteria:

1. Patients with other malignant tumors.
2. Patients with known or suspected autoimmune diseases, including dementia and epilepsy.
3. Patients with severe mental illness.
4. Patients with necrotic lesions and who are assessed by the researchers to be at risk of major bleeding.
5. Patients with severe heart disease, pulmonary dysfunction, heart function and pulmonary function below grade 3 (including grade 3).
6. Patients whose laboratory test values do not meet the relevant standards within 7 days before enrollment.
7. Patients who have received systemic or local glucocorticoid treatment within 4 weeks before enrollment.
8. Patients with complications that require long-term use of immunosuppressive drugs or systemic or local use of corticosteroids with immunosuppressive effects.
9. Patients with active pulmonary tuberculosis (TB) who are currently receiving anti-tuberculosis treatment or have received anti-tuberculosis treatment within 1 year before screening.
10. Previous use of anti-toripalimab, anti-PD-L1 antibody, anti-PD-L2 antibody or anti-CTLA-4 antibody (or any other antibody acting on T cell co-stimulation or checkpoint pathway).
11. Subjects with any active autoimmune disease or history of autoimmune disease (including but not limited to: interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, nephritis, hyperthyroidism, hypothyroidism; patients with vitiligo or complete remission of asthma in childhood and no need for any intervention as adults can be included; patients with asthma requiring medical intervention with bronchodilators cannot be included).
12. HIV positive.
13. HBsAg positive and HBVDNA copy number positive (quantitative detection ≥1000cps/ml); positive blood screening for chronic hepatitis C (HCV antibody positive).
14. Any anti-infection vaccine (such as influenza vaccine, varicella vaccine, etc.) received within 4 weeks before enrollment.
15. Women of childbearing age with positive pregnancy test and breastfeeding women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-06 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) | 2 weeks after the surgery
  pathological complete response rate after radical resection

SECONDARY OUTCOMES:
Major Pathological Response (MPR) | 2 weeks after the surgery
  The proportion of patients whose microscopic tumor cells were reduced to less than 10% as assessed by the American Joint Committee on Cancer/College of American Pathologists (AJCC/CAP) tumor regression grade (TRG) scheme for surgical specimens.
Objective response rate (ORR) | two weeks after the chemoimmunotherapy
  The proportion of patients with a 30% reduction in tumor volume is the sum of the complete response (CR) and partial response (PR) rates.
Disease-free survival (DFS): | 2 years
  The interval from the start of treatment to the earliest treatment failure due to any reason (including local recurrence, regional recurrence, distant metastasis, or death).
Overall survival (OS) | 2 years
  the time interval from the start of treatment to death from any cause.
Mandibular preservation rate: | immediately after the surgery
  the proportion of patients with oral cancer whose mandibular continuity is preserved after primary lesion surgery.
Incidence of adverse events (AEs) and serious adverse events (SAEs) | one month after the postoperative radiotherapy
  the proportion of patients with adverse events of grade 3 or above among all patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiation Oncology, Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) might not be shared due to concerns about patient privacy, ethical considerations, or institutional policies. Restrictions may also arise from data protection regulations, confidentiality agreements, or the potential risk of re-identification. Additionally, if the data includes sensitive medical information, sharing may require special approvals or de-identification processes that are not feasible.

REFERENCES:
- [Background] Caudell JJ, Gillison ML, Maghami E, Spencer S, Pfister DG, Adkins D, Birkeland AC, Brizel DM, Busse PM, Cmelak AJ, Colevas AD, Eisele DW, Galloway T, Geiger JL, Haddad RI, Hicks WL, Hitchcock YJ, Jimeno A, Leizman D, Mell LK, Mittal BB, Pinto HA, Rocco JW, Rodriguez CP, Savvides PS, Schwartz D, Shah JP, Sher D, St John M, Weber RS, Weinstein G, Worden F, Yang Bruce J, Yom SS, Zhen W, Burns JL, Darlow SD. NCCN Guidelines(R) Insights: Head and Neck Cancers, Version 1.2022. J Natl Compr Canc Netw. 2022 Mar;20(3):224-234. doi: 10.6004/jnccn.2022.0016. PMID 35276673
- [Background] Harrington KJ, Burtness B, Greil R, Soulieres D, Tahara M, de Castro G Jr, Psyrri A, Brana I, Baste N, Neupane P, Bratland A, Fuereder T, Hughes BGM, Mesia R, Ngamphaiboon N, Rordorf T, Wan Ishak WZ, Lin J, Gumuscu B, Swaby RF, Rischin D. Pembrolizumab With or Without Chemotherapy in Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma: Updated Results of the Phase III KEYNOTE-048 Study. J Clin Oncol. 2023 Feb 1;41(4):790-802. doi: 10.1200/JCO.21.02508. Epub 2022 Oct 11. PMID 36219809
- [Background] Noronha V, Goswami C, Patil S, Joshi A, Patil VM, Murthy V, Arya S, Juvekar S, Goud S, Prabhash K. Response to docetaxel and cisplatin induction chemotherapy of locally advanced head and neck squamous cell carcinoma: a multicenter, non-comparative, open-label interventional pilot study. J Laryngol Otol. 2016 Sep;130(9):833-42. doi: 10.1017/S0022215116008513. Epub 2016 Jul 26. PMID 27456399
- [Background] Herman LC, Chen L, Garnett A, Feldman LE, Smith B, Weichselbaum RR, Spiotto MT. Comparison of carboplatin-paclitaxel to docetaxel-cisplatin-5-flurouracil induction chemotherapy followed by concurrent chemoradiation for locally advanced head and neck cancer. Oral Oncol. 2014 Jan;50(1):52-8. doi: 10.1016/j.oraloncology.2013.08.007. Epub 2013 Sep 19. PMID 24055193
- [Background] Forastiere AA, Zhang Q, Weber RS, Maor MH, Goepfert H, Pajak TF, Morrison W, Glisson B, Trotti A, Ridge JA, Thorstad W, Wagner H, Ensley JF, Cooper JS. Long-term results of RTOG 91-11: a comparison of three nonsurgical treatment strategies to preserve the larynx in patients with locally advanced larynx cancer. J Clin Oncol. 2013 Mar 1;31(7):845-52. doi: 10.1200/JCO.2012.43.6097. Epub 2012 Nov 26. PMID 23182993
- [Background] Choi YJ, Chung J, Shin HJ, Cho GJ, Wang SG, Lee BJ, Cho BM, Kim DW, Kim HJ, Lee WS, Joo YD, Sohn CH. Induction chemotherapy of docetaxel and Cisplatin for the elderly patients with squamous cell carcinoma of the head and neck. Cancer Res Treat. 2007 Mar;39(1):1-5. doi: 10.4143/crt.2007.39.1.1. Epub 2007 Mar 31. PMID 19746234
- [Background] Lorch JH, Goloubeva O, Haddad RI, Cullen K, Sarlis N, Tishler R, Tan M, Fasciano J, Sammartino DE, Posner MR; TAX 324 Study Group. Induction chemotherapy with cisplatin and fluorouracil alone or in combination with docetaxel in locally advanced squamous-cell cancer of the head and neck: long-term results of the TAX 324 randomised phase 3 trial. Lancet Oncol. 2011 Feb;12(2):153-9. doi: 10.1016/S1470-2045(10)70279-5. Epub 2011 Jan 11. PMID 21233014
- [Background] Vermorken JB, Remenar E, van Herpen C, Gorlia T, Mesia R, Degardin M, Stewart JS, Jelic S, Betka J, Preiss JH, van den Weyngaert D, Awada A, Cupissol D, Kienzer HR, Rey A, Desaunois I, Bernier J, Lefebvre JL; EORTC 24971/TAX 323 Study Group. Cisplatin, fluorouracil, and docetaxel in unresectable head and neck cancer. N Engl J Med. 2007 Oct 25;357(17):1695-704. doi: 10.1056/NEJMoa071028. PMID 17960012
- [Background] Chow LQM. Head and Neck Cancer. N Engl J Med. 2020 Jan 2;382(1):60-72. doi: 10.1056/NEJMra1715715. No abstract available. PMID 31893516
- [Background] Siegel RL, Miller KD, Wagle NS, Jemal A. Cancer statistics, 2023. CA Cancer J Clin. 2023 Jan;73(1):17-48. doi: 10.3322/caac.21763. PMID 36633525